CLINICAL TRIAL: NCT05109611
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled, Phase 3 Clinical Efficacy Study Evaluating Nitric Oxide Nasal Spray (NONS) as Prevention for Treatment of Individuals at Risk of Exposure to COVID-19 Infection
Brief Title: Nitric Oxide Nasal Spray (NONS) as Prevention for Treatment of Individuals at Risk of Exposure to COVID-19 Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment challenges, i.e., not able to meet sample size targeted; secondary to the changing landscape of COVID-19 infection pathology.
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVID-NONS-04
Record Dates: First submitted 2021-11-03; First posted 2021-11-05 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Nitric Oxide; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical labeled nasal spray bottles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide Releasing Solution (Active Comparator): Nasal spray with nitric oxide releasing solution (NORS) delivered up to 3 times daily morning, mid-day, and evening.
  Maximum volume delivered: 0.56 mL NORS @ 0.11ppm*hrs
  Interventions: Drug: Nitric Oxide
- Placebo (Placebo Comparator): Nasal spray with isotonic saline delivered up to 3 times daily morning, mid-day, and evening.
  Maximum volume delivered: 0.56 mL Saline @ 0.9%
  Interventions: Device: Nasal spray with isotonic saline

INTERVENTIONS:
Drug: Nitric Oxide — The Sponsor designed a dual chamber nasal spray bottle for NORS administration. Components are mixed from two chambers to create the final NO-producing formulation. The liquid contains NO at 0.11 ppm*hour, which acts as a viricidal agent. Instructions for storing, preparing, and administering the study treatment will be provided to participants.
  Other Names: Nasal Spray
  Arms: Nitric Oxide Releasing Solution
Device: Nasal spray with isotonic saline — The Sponsor designed a dual chamber nasal spray bottle for NORS administration. The bottle will be filled with normal saline before being provided to the participant.
  Other Names: Normal saline, 0.9% saline
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blinded, placebo-controlled, phase 3 clinical efficacy study evaluating nitric oxide nasal spray (NONS) as prevention for treatment of individuals at risk of exposure to COVID-19 infection.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, placebo-controlled, Phase 3 clinical efficacy study evaluating NONS in adult volunteers as a prevention treatment for individuals at risk from COVID-19 infection.

Up to 13 000 adult participants aged 18 or over with no known history of SARS-CoV-2 infection will be randomized into one of 2 cohorts of this study in a ratio of 1:1 (Treatment: Placebo Control). Participants with or without underlying medical conditions will be eligible to enroll. The NONS formulation proposed for use in this COVID-19 clinical study will be self-administered at a maximum of 3 times per day, morning, noon, and night for 28 days. Participants will be on study for 4 weeks of treatment (to include 5 days of Screening, 1 week of Follow-Up, participants will be followed for a total of approximately 5 weeks) as a viricidal Investigational Medical Product.

Participants will self-administer a nasal spray containing either blinded study treatment or placebo (herein called study treatment). Nitric oxide nasal spray will be delivered from manual pump nasal spray container with 25 mL of solution with each nasal spray dispensing approximately 130-150 µL of solution. After the participant blows their nose, each treatment will require 2 sprays per nostril, or about 0.5 mL per treatment.

The primary endpoint is to assess the efficacy of NONS in the prevention of symptomatic COVID-19 infection as determined by a positive COVID-19 test (antigen or reverse-transcriptase polymerase chain reaction [RT-PCR]),

ELIGIBILITY:
Inclusion Criteria Each participant must meet the following criteria to be enrolled in this study.

1. At least aged 18 years old at the time of consent.
2. If female, be surgically sterile or post-menopausal (no menses for at least 12 months), or if of childbearing potential, must be using an acceptable method of contraception such as a combination estrogen/progestin hormonal contraceptive (oral or injected) for at least 1 month prior to Day 1, or such items as an IUD, intrauterine system (IUS), transdermal hormonal implant, vaginal hormonal ring, or 2 forms of the following: diaphragm, cervical cap, patch, condom, spermicide, or sponge. Total abstinence is permitted. If local regulations deviate from the previously listed contraception methods to prevent pregnancy, local requirements will apply. In addition, females of childbearing potential must agree to continue to use their method of birth control for the duration of the study and 12 weeks following discharge from the study.
3. If male, be surgically sterile, or agree to use appropriate contraception (latex condom with spermicide) when engaging in sexual activity and agree to not donate sperm for the duration of the study and 12 weeks following discharge from the study.
4. Be in good health (ie, no acute illnesses or hospitalizations within 30 days of the study start, no planned procedures during study participation, and no newly diagnosed chronic illnesses that are not deemed stable by the participant's primary care physician), in the opinion of the Investigator, based on medical history (ie, absence of any clinically relevant abnormality) during Screening.
5. Be able to understand and provide written, informed consent.
6. Access to a telephone, the internet, a device that reliability connects to the internet, and able to dial into telehealth checkups and study-related assessments. If access to the internet precludes involvement, then paper diaries may be completed and promptly entered into the data capture system at the study centers as part of the regular follow-up visits.
7. Must be able to receive study product shipments directly to their home (ie, no Post Office Boxes), unless in a region (EU) or other location where the participant must receive the study product directly from the sites' staff/physician.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from the study.

1. Participants with acute illnesses or hospitalizations within 30 days of the study start, and/or planned procedures during study participation, and/or newly diagnosed chronic illnesses that are not deemed stable by the participant's primary care physician), based on Investigator assessment of medical history during Screening.
2. Participants with any respiratory infection, flu-like symptoms, or unexplained fever or chills during the week prior to Screening (see Section 6.6.2).
3. Participants with any prior history of SARS-CoV-2 infection.
4. Participants who use intranasally dosed drugs, prescriptions or over-the-counter medications such as fluticasone within the last 7 days.
5. Participants who underwent a previous tracheostomy.
6. Participants who are receiving any form of oxygen therapy.
7. Females who are breastfeeding, pregnant, or attempting to become pregnant.
8. Participants who have any other condition that, in the opinion of the Investigator, would interfere with a participant's ability to adhere to the protocol (eg, participants whom are mentally or neurologically disabled and whom are considered not fit to their participation in the study), interfere with assessment of the investigational product, or compromise the safety of the participant or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1389 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Moore, PHARMD, Study Director — Sanotize Research and Development corp.
Locations (6):
- Medical Trust Clinics , Inc, Oshawa, Ontario, Canada
- Sri Lanka (5):
  - National Institute of Infectious Diseases Hospital, Angoda, Angoda
  - Karapitiya teaching Hospital,, Galle
  - Peradeniya Teaching Hospital,, Peradeniya
  - Puttalam Base Hospital,, Puttalam
  - Colombo North Teaching Hospital,, Ragama

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1393 participants screened; 1389 participants randomized, 4 screen failures due to participants' having a prior history of SARS-CoV-2 infection.
Groups:
- Nitric Oxide Nasal Spray (NONS): Participants received NONS for 28 days. 695 participants were randomized, 690 participants received at least one dose. 671 (96.5%) participants were compliant with daily use of therapy.
- Saline Nasal Spray (PLACEBO): Participants received PLACEBO for 28 days. 694 participants were randomized, 694 participants received at least one dose. 676 (97.4%) participants were compliant with daily use of therapy.
Period: Overall Study
Arm/Group | Nitric Oxide Nasal Spray (NONS) | Saline Nasal Spray (PLACEBO)
Started | 690 (695 participants randomized; 5 participants did not receive a dose.) | 694
Completed | 674 (690 completed per mITT and used in the safety analysis population, 674 completed PP.) | 677 (694 completed per mITT and used in the safety analysis population. 677 completed PP.)
Not Completed | 16 | 17
Not completed — Adverse Event | 13 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 0 | 4
Not completed — Information unavailable | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants received 3 doses (2 sprays [approx. 0.130 mL/spray] per nostril, max 0.560 mL total/dose) for 28 days. Subjects considered COVID-19 infection-free at randomization. Clinical infection development assessed by nasal swabs and disease severity, i.e., systemic involvement including fever, fatigue, shortness of breath, cough, muscle body aches, nausea, vomiting, diarrhea and nasal/throat symptoms.
Groups:
- Intervention: Nitric oxide nasal spray (NONS)
- Control: 0.9% Sodium chloride nasal spray
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 690 | 694 | 1384
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 667 | 668 | 1335
  >=65 years | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (13.90) | 39.5 (13.68) | 40.0 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364 | 354 | 718
  Male | 326 | 340 | 666
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 689 | 692 | 1381
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 651 | 652 | 1303
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 34 | 35 | 69
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a COVID-19 Infection.
Description: Confirmed positive COVID-19 test (Both antigen and SARS-CoV-2 RT-PCR acceptable) by Day 28.
Time Frame: 28 days
Population: All evaluable participants randomized who received at least one dose of the test article (NONS or placebo; mITT) analyzed through the end of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Nitric Oxide Releasing Solution: Nasal spray with nitric oxide releasing solution (NORS) delivered up to 3 times daily morning, mid-day, and evening; 0.5 mL/dose.
- Placebo: Nasal spray with isotonic saline delivered up to 3 times daily morning, mid-day, and evening; 0.5 mL/dose.
Arm/Group | Nitric Oxide Releasing Solution | Placebo
Number analyzed (Participants) | 690 | 694
Participants | 2 | 2

2. Secondary Outcome: Number of Participants Requiring Medical Services.
Description: Hospitalization or ER/ED visits for COVID-19/flu-like symptoms by Day 28.
Time Frame: 28 days
Population: All randomized participants who received at least 1 dose of study intervention (Safety Population)
Measure: Number; unit: participants
Arm/Group | Nitric Oxide Releasing Solution | Placebo
Number analyzed (Participants) | 690 | 694
participants | 1 | 0

3. Secondary Outcome: Number of Participants Reporting Safety Concerns.
Description: Adverse events captured during treatment (i.e., systemic and local nasal/throat events [emphasis on respiratory and nervous system disorders]).
Time Frame: 28 days
Population: All randomized participants who received at least 1 dose of study intervention (Safety Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide Releasing Solution | Placebo
Number analyzed (Participants) | 690 | 694
Participants | 129 | 130

ADVERSE EVENTS:
Time Frame: 35 days.
Groups:
- Nitric Oxide Releasing Solution: Nasal spray with nitric oxide releasing solution (NORS) delivered up to 3 times daily morning, mid-day, and evening.
  Maximum volume delivered: 0.56 mL NORS @ 0.11ppm*hrs
  13 (1.9%) Participants ET due to AEs
- Placebo: Nasal spray with isotonic saline delivered up to 3 times daily morning, mid-day, and evening.
  Maximum volume delivered: 0.56 mL Saline @ 0.9%
  10 (1.4%) Participants ET due to AEs
Arm/Group | Nitric Oxide Releasing Solution | Placebo
All-Cause Mortality (participants affected / at risk) | 0/690 | 0/694
Serious Adverse Events (participants affected / at risk) | 1/690 | 0/694
Other Adverse Events (participants affected / at risk) | 129/690 | 130/694
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitric Oxide Releasing Solution (N=690) | Placebo (N=694)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) — Secondary to COVID-19 Management (mild [Grade 1] severity, considered not related)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitric Oxide Releasing Solution (N=690) | Placebo (N=694)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 52 (52) | 62 (62)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 34 (34)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 23 (23)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 22 (22)
Headache (Nervous system disorders) | 40 (40) | 69 (69)

LIMITATIONS AND CAVEATS:
Safety Population data provided (up to early termination of the study). Study terminated early secondary to changing SARS-CoV-2 pathology; unable to meet total sample size to reach targeted number of event to maintain 90% power for COVID-19 incidence rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT05109611/Prot_SAP_000.pdf